CLINICAL TRIAL: NCT05736055
Title: Validation Of Cambodia Version of Five Minutes Hearing Test to Screening Hearing Loss
Brief Title: Validation Of Cambodia Version of Five Minutes Hearing Test
Acronym: CAM-FMHT
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Dawin Rotha, MD, Principal Investigator, Khon Kaen University
Other Study IDs: 029NECHR
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cambodia Version Five Minutes Hearing Test — The FMHT was developed by American Academy of Otolaryngology-Head and Neck Surgery (AAO-HNS). The FMHT is composed of 15 questions. Each answer is scored as 0, 1, 2 or 3 according to the frequency of experience. If they answered 'never', the score was 0. The answer 'occasionally' scored 1, the answer 'half the time' scored 2, and the answer 'almost always' scored 3. Furthermore, it has shown more aspects, more reliability, and more assessments of the hearing impairment of the patients. is a standard hearing questionnaire. So, we plan to translate the FMHT into Cambodian language and validate by comparing its result with those of audiometry.
  Other Names: CAM-FMHT

SUMMARY:
Seek the simple tool as questionnaire for screening hearing loss. The FMHT was developed by American Academy of Otolaryngology-Head and Neck Surgery (AAO-HNS). It is a standard hearing questionnaire. So, we plan to translate the FMHT into Cambodian language and validate by comparing its result with those of audiometry.

DETAILED DESCRIPTION:
Primary Objective:

To assess sensitivity of the FMHT in Cambodia version (CAM-FMHT) compared with the standard audiometry

Secondary Objective: To assess

1. Specificity of the FMHT in Cambodia version (CAM-FMHT) compared with the standard audiometry
2. Likelihood ratio of the FMHT in Cambodia version (CAM-FMHT) compared with the standard audiometry
3. Predictive value of the FMHT in Cambodia version (CAM-FMHT) compared with the standard audiometry

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years old
* Able to read and understand Khmer language
* Volunteer to participated

Exclusion Criteria:

* Aphasia patients
* Patients with severe mental disability
* Patients with other conditions that preclude audiometry

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The Cambodian patients complained about hearing problems. They undergo check with audiometry in Preah Ang Duong Hospital, Phanom Penh, Cambodia
Sampling Method: Non-Probability Sample
Enrollment: 481 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
sensitivity of the questionnaire (FMHT in Cambodia version (CAM-FMHT)) | 2 years
  The questionnaire will be used to measure the outcome (score 0 (better outcome)-score45 (worse outcome))

SECONDARY OUTCOMES:
specificity of the questionnnaire (FMHT in Cambodia version (CAM-FMHT)) | 2 years
  The questionnaire will be used to measure the outcome (score 0 (better outcome)-score45 (worse outcome))
likelihood ratio of the questionnaire (FMHT in Cambodia version (CAM-FMHT)) | 2 years
  The questionnaire will be used to measure the outcome (score 0 (better outcome)-score45 (worse outcome))
predictive value of the questionnaire (FMHT in Cambodia version (CAM-FMHT)) | 2 years
  The questionnaire will be used to measure the outcome (score 0 (better outcome)-score45 (worse outcome))

CONTACTS AND LOCATIONS:
Overall Officials: Dawin Rotha, M.D., Principal Investigator — Khon Kaen University
Locations (1):
- Preah Ang Duong Hospital, Phnom Penh, Cambodia

IPD SHARING:
Plan to Share IPD: No